CLINICAL TRIAL: NCT03749122
Title: Preoperative Waiting Time to Surgery Related to Mortality in Hip Fracture Patients
Brief Title: Time to Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgård, Associate professor, Sahlgrenska University Hospital
Other Study IDs: 331-16
Record Dates: First submitted 2018-11-15; First posted 2018-11-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Hip Fractures; Mortality; Surgery
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Waiting time for hip fracture surgery — Time from hospital admission to start of hip fracture surgery

SUMMARY:
The purpose of the study is to evaluate how time from hospital admission to start of surgery influence mortality in patients with acute hip fracture. Data on patients with hip fracture surgery will be collected from the hospital's registration system and will be analyzed regarding age, gender, American Society of Anesthesiologists (ASA) Physical Status Classification, type of surgery and time from admission to surgery along with data on mortality.

ELIGIBILITY:
Inclusion Criteria: undergoing

* hip fracture surgery between 2007-2016.
* Over 60 years of age.

Exclusion Criteria:

* Pathological fracture.
* In-hospital falls.
* Diagnostic delay.

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Date of Death captured through Swedish Taxation Authority within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Bengt, Mölndal, V. Götaland, Sweden

IPD SHARING:
Plan to Share IPD: No